CLINICAL TRIAL: NCT05058508
Title: LCI-PED-NOS-EXER-001: Just Move. A Randomized Controlled Trial Investigating Exercise in Pediatric Oncology Patients
Brief Title: LCI-PED-NOS-EXER-001: Exercise in Pediatric Oncology Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00082746; LCI-PED-NOS-EXER-001 (Other: Atrium)
Record Dates: First submitted 2021-09-14; First posted 2021-09-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Cancer
Keywords: Exercise; Pediatric Oncology
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXER (Experimental): "Just Move" exercises
  Interventions: Other: "Just Move" Exercise
- SOC EXER (Experimental): Standard of Care Exercise
  Interventions: Other: Standard of Care Exercise

INTERVENTIONS:
Other: "Just Move" Exercise — Subjects complete "Just Move" Exercises Five Times Per Week
  Arms: EXER
Other: Standard of Care Exercise — Subjects exercise/move as tolerated
  Arms: SOC EXER

SUMMARY:
The purpose of this study is to see if there are physical and emotional benefits to participating in a structured exercise regimen for those who are ages 2-25, are newly diagnosed with a blood or solid tumor cancer, and are currently undergoing or will begin cancer treatment.

DETAILED DESCRIPTION:
This is a randomized, controlled trial to investigate if a structured exercise regimen will have benefit relative to the control arm by increasing and /or maintaining physical functioning in pediatric subjects undergoing chemotherapy and childhood cancer treatment as measured by 6-Minute Walk test and BOT-2 Brief or PDMS-2.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 2-25 at time of consent
2. Subject has newly diagnosed cancer per Investigator, and is planning to undergo chemotherapy for treatment of malignancy for at least 3 full cycles
3. Ability of subject (and/or parent/guardian) to read and understand the English or Spanish language
4. As determined and documented by the enrolling investigator, ability of the subject to understand and comply with study procedures for the entire length of the study
5. Subject has newly diagnosed cancer per Investigator and is planning to undergo chemotherapy, immunotherapy, or other systemically delivered for treatment of malignancy. Subjects are allowed to be enrolled up to 21 days after initiating cancer treatment.
6. Receiving oncologic care at Levine Children's Cancer and Blood Disorders Clinic.
7. Subject is anticipated to receive at least 3 full cycles of chemotherapy or other systemic cancer treatment.
8. Not participating in another clinical trial that precludes participating in additional nondrug clinical trials.

Exclusion Criteria:

1. Known cardiac dysfunction that, in the opinion of the investigator, would be unsafe for the child to participate in the exercise program
2. Any other uncontrolled intercurrent illness/medical condition or psychiatric illness/social situations that would limit compliance with study requirements or would be considered unsafe for the child to participate as determined by the Investigator.
3. Recent (within 4 weeks of enrollment) or planned surgery that will result in prolonged limited mobility not amendable to exercise modifications per investigator discretion
4. Primary CNS Tumor
5. Osteosarcoma

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Potential benefit of increasing/maintaining physical functioning in pediatric subjects undergoing chemotherapy and childhood cancer treatment | 18 month period
  Investigate if 30 minutes of exercise, five days per week, will have benefit relative to the control arm by increasing and/or maintaining physical functioning in pediatric subjects undergoing chemotherapy and childhood cancer treatment as measured by 6-Minute Walk test
Potential benefit of increasing/maintaining physical functioning in pediatric subjects undergoing chemotherapy and childhood cancer treatment | 18 month period
  Investigate if 30 minutes of exercise, five days per week, will have benefit relative to the control arm by increasing and/or maintaining physical functioning in pediatric subjects undergoing chemotherapy and childhood cancer treatment as measured by BOT-2 Brief (in subjects ≥ 4 years of age) or PDMS-2 (in subjects < 4 years of age).

SECONDARY OUTCOMES:
Adverse Event Rate | up to 18 months
  Occurrence of Adverse Events of Special Interest (thromboembolic event, skin ulceration, significant nausea/vomiting, and constipation) will be measured as binary variables.
Quality of Life measured by the PedsQL Cancer Module | up to 18 months
  Investigate if a structured exercise regimen relative to the control arm will result in Increasing and /or maintaining quality of life as measured by the PedsQL Cancer Module. Peds QL scores will be calculated as a composite quantitative analogue variable ranging from zero (best score) to 100 (worst score).
Subject adherence to exercise regimen | up to 18 months
  Subject adherence to exercise regimen will be determined by patient-reported tracker listing activity performed and duration of time of activity. Data collected will be normalized quantitatively based on intended activity.
Adverse Events Related to Exercise Program | up to 18 months
  To summarize adverse event rates deemed to be related to the protocol directed exercise program. Adverse events of special interest (Grade 2 or greater Bone fracture, Fall, and Muscle aches/Myalgia) will be captured for each subject and time point randomized to the intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Pope, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Children's Hospital, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No